CLINICAL TRIAL: NCT05619835
Title: A Usability Study of a Tele-health Service for Patients With Peripheral Arterial Disease.
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: AIT Austrian Institute of Technology GmbH (Other)
Responsible Party: Principal Investigator, Günther Silbernagel, Assoc.-Prof. Priv.-Doz. Dr.med.univ. et scient.med., Medical University of Graz
Other Study IDs: 1566-2021
Record Dates: First submitted 2022-05-07; First posted 2022-11-17 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Walking exercise; Tele-health Service; Disease Management Program; Preventive Medicine; Integrated care; Vascular Medicine
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to analyze the applicability (usability) of a tele-health service as part of a potential disease management program for patients with peripheral arterial disease.

The following investigations will be conducted as part of the usability study. In the context of a tele-health service, knowledge, physical condition (including walking distance) will be documented during face-to-face and televisits, dislocated supervised gait training and education will be provided, and satisfaction with the tele-health service will be evaluated.

DETAILED DESCRIPTION:
Disease management programs (DMPs) are one of the methods used to optimize the care of patients with chronic diseases. DMPs are coordinated health care measures for patient populations with diseases in which active patient participation in treatment can lead to substantial effects. Specific treatment regimens, based on evidence-based treatment guidelines and structured patient information, are predominantly aimed at preventing disease exacerbations and complications. The World Health Organization (WHO) also recommends, among other things, forcing patient adherence through structured information and patient empowerment strategies to establish participatory treatment.

Peripheral arterial disease (PAD) causes oxygen and nutrient deprivation of tissues through narrowing of arterial vessels in the extremities. The cause of PAD is arteriosclerosis. The course of the disease begins asymptomatically and manifests itself over time with pain and cramps predominantly in the muscles of the lower extremity. The pain symptoms usually occur initially during physical exertion, and later at rest. As PAD progresses, chronic ulceration and necrosis occur.

Professional societies such as the European Society of Cardiology (ESC) and the European Society of Vascular Medicine (ESVM) regularly publish guidelines for the diagnosis and treatment of PAD. Therapy of PAD consists of drug therapy for the purpose of cardiovascular risk reduction (lipid and blood pressure lowering drugs and anticoagulant drugs as well as therapy of diabetes mellitus). Another aspect in the event of disease progression is interventional angioplasty, in which the affected constriction in the leg arteries is dilated and, if necessary, treated with stents. Another important pillar is also structured and supervised gait training and, in general, an improvement in lifestyle with cessation of nicotine abuse and a healthy diet.

In particular, structured gait training, which should be performed at least three times a week for 30 to 60 minutes, is strongly recommended in the current ESVM and ESV guidelines. Studies showed that structured gait training can increase walking distance by 200% in 12 weeks in patients with claudication. Daily individual interval training of 60 minutes with 5- to 15-minute intervals also proved effective in increasing walking distance. This is to overcome the pain threshold of claudication while walking. Furthermore, evidence showed that gait training may be equivalent to endovascular interventions in terms of long-term outcomes.

The aim of this study is to analyze the applicability (usability) of a telehealth service as part of a potential disease management program for patients with peripheral arterial disease.

A prospective monocentric pilot study will be conducted at the clinical department of angiology.

The study duration per participant is 90 (±14) days and is divided into 2 observation phases. In phase 1, there will be supervision by a certified nurse and the telehealth service app, and in phase 2, there will be only singular use of the app without contact by the certified nurse.

The Declaration of Helsinki (as amended from time to time) and the guidelines of "Good Clinical Practice" were taken into account in the conduct and also the planning of the study.

Furthermore, the framework guideline for the "IT infrastructure in the application of telemonitoring" was used for the planning of the study.

According to the manufacturer's manuals, the pedometers AS80/AS97/AS99 from the company Beurer are not medical devices. The app serves as a diary for patients and is not a Clinical Decision Support System. The "User's Manual PAD Stepping" is included with the study material.

Reference Projects:

The DMS app system is also already being used in routine care in the "Herzmobil" project in Styria and Tyrol. Here, patients with chronic heart failure are cared for.

The use of the DMS app is currently also being used in two other studies. These are observational studies that are not subject to the Medical Devices Act. Both projects have a positive ethics vote and are listed under the following titles:

* Telemedical follow-up of hospitalized patients with coronavirus disease-2019 (COVID-19) DRKS ID of the study: DRKS00022244.
* Building a training database of voice data recordings and body weight trajectories in hemodialysis patients for algorithm development.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of "peripheral arterial occlusive disease" in, IIa and IIb (according to Fontaine).
* Age between 18 and 80 years
* Written informed consent
* Smartphone with Android operating system
* Understanding of how to use the tele-health service

Exclusion Criteria:

* Patients with PAD stages I, III and IV (according to Fontaine)
* Lack of compliance
* Smartphone with non-Android operating system or incompatible software

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with IIa and IIb PAD at the Department of Angiology at the LKH-University Hospital Graz.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with the telehealth service. | At time point visit 3, which is 12 weeks after baseline
  Study participants will undergo guided interviews measuring patient satisfaction with telehealth service.

SECONDARY OUTCOMES:
Proportion of patients, who would be satisfied with the telehealth service if telephone calls would not be provided by a nurse during the programme | At time point visit 3, which is 12 weeks after baseline
  Yes/No
Change of walking distances in the 6 minute walk test determined by the certified nursing staff in response to the telehealth service. | From baseline to visit 3, which is 12 weeks after baseline
  Walking distances in the 6 minute walk test will be determined by the certified nursing staff.
Change of subjective limitations in the activities of daily living. | From baseline to visit 3, which is 12 weeks after baseline
  Study participants will undergo a questionaire (SF36) measuring subjective limitations in the activities of daily living.
Change of knowledge about peripheral arterial disease. | From baseline to visit 3, which is 12 weeks after baseline
  Study participants will undergo a questionaire measuring knowledge about peripheral arterial disease before and 12 weeks after a structured education.
Total number of performed 6 minute walk tests during the telehealth service. | At time point visit 3, which is 12 weeks after baseline
  Study participants will perform 6 minute walk tests independently using the App during the telehealth service.
Differences of the walking distance in the same 6 minute walk test determined by the nursing staff compared the App. | At baseline and at visit 3, which is 12 weeks after baseline
  Walking distances in the 6 minute walk test will be determined by the certified nursing staff as well as by the App.
Average steps per day during the telehealth service. | From baseline to visit 3, which is 12 weeks after baseline
  Descriptive
Change of summed seconds in the "Time up and Go Test". | From baseline to visit 3, which is 12 weeks after baseline
  The "Time up and Go Test" will be performed by an installed automatic measure system and will be observed by the certified nursing staff. The patient has to stand up from a chair and walk three meter straight. The time needed for this procedure will be measured exactly by a sensor supported measure system.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided